CLINICAL TRIAL: NCT00130819
Title: Buprenorphine Effectiveness Evaluation in HIV Enhancement (BEEHIVE): A Randomized Trial of HIV Clinic-based Buprenorphine/Naloxone vs. Case Management and Referral in Opioid-dependent Individuals
Brief Title: Comparison of HIV Clinic-based Treatment With Buprenorphine Versus Referred Care in Heroin-dependent Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The New York Academy of Medicine (Other)
Responsible Party: Gregory M. Lucas, MD PhD, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H97HA03794; HRSA-04-078
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Opiate Dependence; HIV Seropositivity; HIV Infections
Keywords: Drug Dependence; Opiate Dependence; Human Immunodeficiency Viruses; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; HIV Seropositivity; HIV Infections; Substance-Related Disorders; Acquired Immunodeficiency Syndrome | interventions — Buprenorphine; Case Management

ARMS (2):
- 1 (Experimental): Subjects receive integrated opioid-dependence treatment with buprenorphine/naloxone at the HIV clinic
  Interventions: Behavioral: Clinic-based substance abuse treatment with buprenorphine
- 2 (Active Comparator): Subjects receive case management and referral to an off-site opioid treatment program for their opioid dependence
  Interventions: Behavioral: Case management and referred substance abuse treatment

INTERVENTIONS:
Behavioral: Clinic-based substance abuse treatment with buprenorphine — Subjects receive integrated opioid-dependence treatment with buprenorphine/naloxone at the HIV clinic
  Arms: 1
Behavioral: Case management and referred substance abuse treatment — Subjects receive case management and referral to an off-site opioid treatment program for their opioid dependence
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of two approaches to treating HIV-infected patients who are addicted to opioid drugs (e.g., heroin) in an inner-city HIV clinic. The two approaches are:

* Case management and referral - participants are managed by a case manager and referred to a specialized drug treatment center where they receive counseling and medications for opioid-dependence (e.g., methadone or buprenorphine); or
* Clinic-based treatment - participants receive counseling and treatment with buprenorphine at the HIV clinic.

DETAILED DESCRIPTION:
We, the investigators at Johns Hopkins University, propose to enroll and randomize 120 opioid-dependent, HIV-infected participants, who receive care in the Johns Hopkins HIV Clinic to either:

* clinic-based care with buprenorphine (clinic-based BPN/NX arm); or
* case management and referral to an opioid treatment program for opioid agonist-based therapy (case management and referral arm).

The study interventions and follow-up will last 12 months. Participants will be enrolled over a 3-year period. Participants who are assigned to the clinic-based BPN/NX arm will receive BPN/NX (Suboxone®), individual counseling from a nurse interventionist, and group therapy sessions. Participants who are assigned to the case management and referral arm will be enrolled in an established case management and adherence program in the Johns Hopkins HIV Clinic (Project LINK). LINK provides intensive case management, education, and support by a team that includes a social worker, a nurse, a pharmacist educator, and peer advocates. In addition to providing counseling and linkage to needed services, LINK will expedite intake at licensed opioid treatment programs that provide agonist-based therapy for opioid dependence. The clinic-based BPN intervention is a new strategy that was developed in a pilot project over the past 6 months. The case-management and referral arm represents standard-of-care in our clinic, which has been enhanced and codified for this trial. Study outcome visits will be performed at baseline, 1 month, 3 months, 6 months, 9 months, and 12 months.

Comparisons:

* Retention to substance abuse treatment;
* Urine drug screens;
* Adherence to HIV primary care provider visits;
* Use of and adherence to highly active antiretroviral therapy (HAART);
* HIV RNA levels and CD4 cell counts;
* HIV transmission risk behaviors (e.g., injection, sharing of drug paraphernalia, sexual behaviors);
* Costs and resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected and receiving continuity care in the Johns Hopkins HIV Clinic
* 18 years of age or older
* Meets DSM-IV criteria for opioid dependence
* Seeks agonist-based treatment for opioid dependence
* Willing and able to provide written informed consent
* Willing to be contacted by mail and telephone for study follow-up visit reminders
* Willing to authorize release of information for substance abuse treatment to the study for a period of 12 months
* If female, negative urine pregnancy test and willingness to practice birth control while on study if sexually active (barrier method or progesterone-containing contraception product)
* Verbal approval from participant's primary HIV clinician

Exclusion Criteria:

* Currently receiving methadone, naloxone, buprenorphine, or levomethadyl acetate (LAAM) as part of a licensed opioid treatment program
* History of allergic reaction to buprenorphine or naloxone
* Active medical need for opioid-based pain control
* Active benzodiazepine abuse or dependence
* Active alcohol dependence
* Alanine aminotransferase level that is more than 5 times the upper limit of normal
* Other condition that, in the opinion of the principal investigator, makes participation in the study unsafe or follow-up highly unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Retention to substance abuse treatment | 12 months

SECONDARY OUTCOMES:
Visit attendance with primary medical provider | 12 months
Urine drug screen positivity for opioids and other drugs | 12 months
Use of and adherence to highly active antiretroviral therapy (HAART) | 12 months
HIV RNA changes | 12 months
CD4 cell count changes | 12 months
Self-reported HIV transmission risk behaviors | 12 months
Costs and resource utilization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Lucas, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins HIV Clinic, Baltimore, Maryland, United States

REFERENCES:
- [Result] Lucas GM, Chaudhry A, Hsu J, Woodson T, Lau B, Olsen Y, Keruly JC, Fiellin DA, Finkelstein R, Barditch-Crovo P, Cook K, Moore RD. Clinic-based treatment of opioid-dependent HIV-infected patients versus referral to an opioid treatment program: A randomized trial. Ann Intern Med. 2010 Jun 1;152(11):704-11. doi: 10.7326/0003-4819-152-11-201006010-00003. PMID 20513828
- See also: Coordinating site webpage — http://www.bhives.org/